CLINICAL TRIAL: NCT07376395
Title: The Effect of Jin Shin Jyutsu-Based Hand Application Guided by the Transactional Model of Stress and Coping on Quality of Life and Psychosocial Status in Perimenopausal Women
Brief Title: Effects of Jin Shin Jyutsu-Based Hand Application on Quality of Life and Psychosocial Status in Perimenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eslem Altıntaş, M.Sc., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-20/740
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Quality of Life; Depression; Anxiety; Stress
Keywords: Perimenopause; Quality of Life; Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jin Shin Jyutsu-Based Hand Application (Experimental): Participants assigned to this arm will receive a Jin Shin Jyutsu®-based hand application intervention guided by the Transactional Model of Stress and Coping. The intervention includes an initial individual training session (approximately 30-40 minutes) providing education on stress, coping, and the principles of Jin Shin Jyutsu®, followed by a structured self-application protocol. Participants will practice the hand application daily for 14 consecutive days, for at least 15 minutes per day, and will be supported with reminder messages to enhance adherence. This intervention is designed as a supportive self-care approach rather than a medical treatment.
  Interventions: Behavioral: Jin Shin Jyutsu®-Based Hand Application
- Control Group (Active Comparator): Participants assigned to this arm will receive standard informational counseling related to general health during perimenopause. This includes a brief verbal education session (approximately 10-15 minutes) covering perimenopause-related changes and general lifestyle recommendations, such as sleep hygiene, balanced nutrition, physical activity, and stress awareness. No Jin Shin Jyutsu® techniques or relaxation interventions will be provided during the study period. Outcome assessments will be conducted at the same time points as the experimental group.
  Interventions: Behavioral: General Health Education

INTERVENTIONS:
Behavioral: General Health Education — Participants assigned to the control group will receive standard verbal health education related to general health during perimenopause. The content includes information on common perimenopausal changes and general lifestyle recommendations. No Jin Shin Jyutsu® techniques, relaxation exercises, or structured coping interventions are included.
  Arms: Control Group
Behavioral: Jin Shin Jyutsu®-Based Hand Application — Participants assigned to the experimental arm will receive a Jin Shin Jyutsu®-based hand application program guided by the Transactional Model of Stress and Coping. During the initial session, participants will receive a structured face-to-face training lasting approximately 30-40 minutes, including verbal instruction, visual materials, and a practical demonstration of the hand application techniques.
  Participants will be instructed to practice the Jin Shin Jyutsu® hand application daily for at least 15 minutes over a 14-day period. The intervention is designed as a self-care-based supportive approach and does not involve medical treatment, physical manipulation, or pharmacological therapy.
  To support adherence, participants will receive written instructions, a daily self-monitoring log, and brief reminder messages via WhatsApp® during the intervention period. No additional therapeutic techniques or relaxation interventions will be provided.
  Arms: Jin Shin Jyutsu-Based Hand Application

SUMMARY:
This study aims to evaluate the effect of Jin Shin Jyutsu-based hand application guided by the Transactional Model of Stress and Coping on quality of life and psychosocial status in perimenopausal women. Participants will receive a structured hand application intervention over a defined period. Outcomes related to quality of life and psychosocial well-being will be assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-54 years
* Being in the perimenopausal period according to the STRAW+10 criteria
* Being literate

Exclusion Criteria:

* Use of hormone replacement therapy
* Regular use of complementary or alternative therapy
* History of diagnosed psychiatric disorders
* Inability to comply with the intervention protocol

Ages: 40 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form | Day 1 (Baseline, Pre-Intervention)
  This is a 24-question form designed by researchers to determine participants' sociodemographic characteristics, women's health status, general health knowledge, lifestyle, and support levels.
Coping Strategies | Day 1 (Baseline, before intervention for intervention groups, before routine assessment for control group) and Day 14 (Post-intervention for intervention groups, after routine assessment for active comparator).
  The Stress Coping Methods Scale (SBÇYÖ) is a self-report questionnaire assessing active and cognitive coping strategies used by adults when facing stressful situations. The scale consists of 21 items rated on a 5-point Likert scale (1-5) and includes five subdomains: logical analysis, positive reappraisal, problem solving, seeking professional support, and seeking environmental support. Total and subscale scores increase as the corresponding coping strategy is used more frequently. Higher scores indicate greater use of the specified coping strategy.
Menopause-Specific Quality of Life | Day 1 (Baseline, before intervention for intervention groups, before routine assessment for control group) and Day 14 (Post-intervention for intervention groups, after routine assessment for active comparator).
  The Menopause-Specific Quality of Life Questionnaire - II (MENQOL / MÖYKÖ-II) is a validated self-report instrument developed to assess the presence and severity of menopause-related symptoms and their impact on quality of life across vasomotor, psychosocial, physical, and sexual domains.
  The scale consists of 29 items. For each item, participants indicate whether the symptom is present; if present, the level of discomfort is rated. Item scores are converted to a 1-8 scoring system. The total score ranges from 29 to 232, with higher scores indicating worse quality of life and greater negative impact of menopausal symptoms.
Distress Thermometer | Day 1 (Baseline, before intervention for intervention groups, before routine assessment for control group) and Day 14 (Post-intervention for intervention groups, after routine assessment for active comparator).
  The Distress Thermometer is a single-item visual analog scale designed to rapidly assess overall psychological distress. Participants rate their distress level on a scale ranging from 0 (no distress) to 10 (extreme distress).
  Higher scores indicate higher levels of psychological distress. In this study, the problem list accompanying the Distress Thermometer is not used.
Depression, Anxiety, and Stress | Day 1 (Baseline, before intervention for intervention groups, before routine assessment for control group) and Day 14 (Post-intervention for intervention groups, after routine assessment for active comparator).
  The Depression Anxiety Stress Scales-21 (DASS-21) is a self-report questionnaire assessing depression, anxiety, and stress symptoms over the past week. It consists of 21 items, with three subscales of seven items each.
  Items are rated on a 4-point Likert scale (0-3). Subscale scores range from 0 to 42 after standard score conversion. Higher scores indicate greater levels of depression, anxiety, and stress, reflecting worse psychological outcomes.
Daily Practice Schedule for JSJ®-Based Hand Application | The intervention group will complete this chart for 14 days.
  This chart, developed by the researchers, is designed for participants to regularly record their daily practices for 14 days. The chart includes the day, total time, whether the five-finger grip was completed, and notes. This chart will be used to monitor the level of adherence to the intervention and the frequency of problem-focused coping actions.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Şahin, Prof. Dr., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Provincial Directorate of Health - Family Health Centers, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No